CLINICAL TRIAL: NCT02443870
Title: Retrospective Analysis of Long-term Urodynamics in Individuals With Neurogenic Lower Urinary Tract Dysfunction
Brief Title: Long-term Urodynamics in Individuals With Neurogenic Lower Urinary Tract Dysfunction
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2013-11
Record Dates: First submitted 2015-05-06; First posted 2015-05-14 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Neurogenic Lower Urinary Tract Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The long-term changes of bladder function in individuals with lower urinary tract dysfunction will be investigated. Patients presenting for regular urodynamic examination of bladder function will be included. Bladder diary details and urodynamic data will be collected in order to investigate bladder function.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic lower urinary tract dysfunction
* urodynamic data

Exclusion Criteria:

* duration of neurogenic lower urinary tract dysfunction < 10 years
* < 5 urodynamic follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with neurogenic lower urinary tract dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
maximal detrusor storage pressure | 12 month after previous investigation

SECONDARY OUTCOMES:
bladder capacity | 12 month after previous investigation
bladder compliance | 12 month after previous investigation
  The relationship between a change in bladder volume and the change in detrusor pressure (ΔDV/ΔDP).
maximal detrusor voiding pressure | 12 month after previous investigation
reflexive bladder volume | 12 month after previous investigation

OTHER OUTCOMES:
gender | time of injury
age | time of injury
lesion level | time of injury
lesion severity | time of injury
bladder evacuation method | 12 month after previous investigation
presence of incontinence | 12 month after previous investigation
complications | 12 month after previous investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland